CLINICAL TRIAL: NCT00429403
Title: Phase III Randomized Study of a Goserelin Acetate for Preservation of Ovarian Function in Patients With Primary Breast Cancer (PBC)
Brief Title: Goserelin Acetate Study for Ovarian Function in Patients With Primary Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0464
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2011-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Chemotherapy; Ovarian Function; Goserelin; Zoladex; Ovary function; Fertility; Early Menopause
MeSH Terms: conditions — Breast Neoplasms; Primary Ovarian Insufficiency | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Goserelin (Experimental): 3.6 mg subcutaneously 1 week before chemotherapy, then once a month until 3 weeks after chemotherapy.
  Interventions: Drug: Goserelin
- No Goserelin (No Intervention)

INTERVENTIONS:
Drug: Goserelin — 3.6 mg subcutaneous injection 1 week before the start of chemotherapy, then once a month until 3 weeks after the last chemotherapy dose.
  Other Names: Zoladex
  Arms: Goserelin

SUMMARY:
Primary Objective:

* To determine the effectiveness of goserelin acetate (Zoladex) in preserving ovarian function in premenopausal women undergoing neoadjuvant and/or adjuvant chemotherapy for primary invasive breast cancer by documenting persistence or resumption of regular menses.

Secondary Objectives:

* To determine the incidence of pregnancy and the effect for participants' quality of life (QOL) after chemotherapy.
* To determine the overall survival and disease-free survival times of study participants.

DETAILED DESCRIPTION:
Goserelin is designed to block hormones that can regulate your menstruation by affecting the pituitary gland (part of brain).

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two treatment groups. You will either be assigned to receive goserelin or no treatment. There is an equal chance of being assigned to either group.

If you are assigned to receive goserelin, the first dose will be given as an injection under the skin, 1 week before you start chemotherapy. You will then receive chemotherapy as part of your standard of care. Following the first dose of goserelin, you will be given a goserelin injection into the skin, once a month until 3 weeks after the last chemotherapy dose.

You will be taken off study if intolerable side effects occur during this study. After you are finished with chemotherapy, you will have a series of follow-up visits. During the period of follow-up, you will have a medical history, physical exam, and blood tests (2-3 teaspoons) to evaluate your ovarian function, every 3 months for 1 year and then at 24 months. You will be asked to fill out questionnaires about your menstrual history at these visits. The questionnaires should take about 15 minutes to complete. You will be also asked to fill out questionnaires about your quality of life at 12 and 24 months. The questionnaires should take about 30 minutes to complete.

This is an investigational study. Goserelin is commercially available and has been approved by the FDA for use in breast cancer patients. Its use in this study is investigational. About 148 patients will take part in this multicenter study. Up to 36 patients will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients older than 15 years and younger than 46 years.
2. Primary breast cancer (Stage I, II, or III).
3. Pathologically confirmed invasive breast carcinoma.
4. Negative hormone-receptor status. (Negative defined as ER- and PR- staining in less than 10% of tumor cells, or tumors with less than or equal to 3 fm/mg cytosol protein on ligand-binding or enzyme-linked immunoassay).
5. Premenopausal, verified before chemotherapy is begun as satisfying both:

   * Cyclic vaginal bleeding.
   * Follicle-stimulating hormone (FSH) is less than or equal to 15 IU/L. If patients are taking oral contraceptives, FSH must be measured 1-2 weeks after discontinuation. If FSH is greater than 15 and the patient has regular menses, gynecologic consultation will be required for a decision on premenopausal status.
6. Candidates for neoadjuvant and/or adjuvant chemotherapy for primary breast cancer.
7. Treatment with at least four (4) cycles of chemotherapy as planned.
8. Zubrod performance score of 0 or 1.
9. Must consent to preservation of their ovarian function and indicate their awareness of the investigational nature of this study, in keeping with institutional policy.
10. Willingness to use barrier contraception if sexually active.

Exclusion Criteria:

1. Pregnancy. Women must have a negative serum pregnancy test before initiation of injection.
2. Hypersensitivity to any GnRH analog.
3. Previous receipt of systemic chemotherapy.
4. To receive at least 4 cycles of neoadjuvant and/or adjuvant chemotherapy with CMF.
5. Stage IV breast cancer.
6. Prothrombin time (PT) and partial prothrombin time (PTT) with INR > 1.5
7. Platelets < 50,000/mm^3

Ages: 15 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2006-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- UT MD Anderson Cancer Center, Houston, Texas, United States
- St. Luke's International Hospital, Tokyo, Japan

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period of Recruitment: August 30, 2006 to August 25, 2009. All patient recruitment made at UT MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early due to slow accrual.
Period: Overall Study
Arm/Group | Goserelin | No Goserelin
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Goserelin | No Goserelin | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Number; unit: years]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response (FSH Level + Vaginal Bleeding)
Description: Outcome characterized in terms of two variables, each measured repeatedly over time: Follicle-stimulating hormone (FSH) level and whether vaginal bleeding occurs, each to be measured from the end of chemotherapy. For treatment comparison, "response" defined as a composite event: both [FSH < 15] and vaginal bleeding observed within 12 months after the end of chemotherapy, with both FSH and vaginal bleeding baseline observed before start of chemotherapy.
Time Frame: Baseline prior to chemotherapy then every 3 months after chemotherapy for 1 year
Population: Analysis was per protocol. Limited analysis due to low recruitment and early termination.
Measure: Number; unit: participants
Arm/Group | Goserelin | No Goserelin
Number analyzed (Participants) | 1 | 0
participants | 1 |

ADVERSE EVENTS:
Time Frame: 2 years and 6 months
Description: There were no participants in the No Goserelin group so the number of participants at risk or affected was null for both serious and/or other [non-serious] adverse events.
Arm/Group | Goserelin | No Goserelin
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No